CLINICAL TRIAL: NCT03375801
Title: Implementing a Decision Aid for Breast Cancer and DCIS Patients Deciding on Their Radiation Treatment: A Pre- and Post-intervention Study.
Brief Title: Implementing a Decision Aid for Breast Cancer and DCIS Patients Deciding on Their Radiation Treatment.
Acronym: BRASA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: M17SDM
Record Dates: First submitted 2017-10-31; First posted 2017-12-18 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: Pre- and post intervention study.
Masking Description: first 164 patients will not receive the decision aid, they will only fill out the questionnaires.
  The next 164 patients will receive the decision aid and will be asked to fill out the same questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group/pre intervention (No Intervention): the first 164 patients will receive care as usual and will make the decision together with their clinician without support of the decision aid. They will be asked to fill out the questionnaires.
- intervention arm (Experimental): another 164 patients will receive the decision aid as support for the decision making process with their clinician.
  Interventions: Other: Decision Aid

INTERVENTIONS:
Other: Decision Aid — This will be an online tool giving evidence based information and explanation on their options.
  Arms: intervention arm

SUMMARY:
This is a pre-and post intervention study on the effect and implementation of an personalized decision aid for woman with breast cancer who face a decision on their radiation treatment.

DETAILED DESCRIPTION:
Rationale: Guidelines on breast cancer treatment show grey areas for some radiotherapy (RT) indications. In some recommendations the uncertainty is marked and deferred to sharing the final decision on the treatment of choice with the patient. Other recommendations are straightforward, but the multidisciplinary team may decide, based on the latest literature, that different options should be discussed with the patient. In these so called "preference sensitive decisions" there is not one best option. The best option depends on the individual patients' preferences based on neutral and complete information tailored to her own situation. Decision aids support clinicians as well as patients in Shared Decision Making (SDM). Decision aids reduce the patient's decisional conflict after making their decision, increase their knowledge on their illness and the treatment options, and their perceived level of involvement in the decision making process. Although extensive research has been carried out on the effect of decision aids in clinical trials, less is known of the effect of a decision aid in daily clinical practice. The implementation of SDM is challenged by many barriers. The investigators hypothesize that adapting the decision aid to individual patient characteristics may enhance both personalised medicine and SDM.

Objective: To investigate whether SDM using a personalised decision aid, results in improved outcomes of decisional quality, measured by the Decisional Conflict Scale after 3 months and one year, and improved outcomes of the decisional process, measured with the SDMQ9 and collaboRATE directly after the last consultation, compared to the standard clinical practices in breast cancer patients facing a decision on their radiation treatment.

Study design: This is a multicenter clustered , pre- and post-intervention study. Before the intervention 164 patients will be included. After introducing the decision aid, at the beginning of the intervention period, clinicians will be trained in using the decision aid and the other 164 patients will be recruited.

Study population: Breast cancer patients facing a decision in their adjuvant radiation treatment.

Intervention: The intervention group will receive the instructions and the online decision aid.

Main study parameters/endpoints: Primary endpoint: Decisional conflict 3 months after the decision has been made. Secondary endpoint(s): The perceived level of shared decision making, patient knowledge, , and decisional conflict 1 year after decision has been made. A process evaluation will also be perform.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Female
* Doubtful indication of:

  * Whole breast irradiation after lumpectomy for DCIS
  * Whole breast irradiation after lumpectomy for low risk invasive BC (TOP-1 study)
  * Boost dose in case of Breast Conserving Therapy
  * Thoracic wall irradiation post mastectomy

Exclusion Criteria:

* Metastasis
* Inability to speak and read Dutch. Inability to use internet access, either in the home or at a hospital facility.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 403 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
Decisional conflict | 90 days after the decision on their radiation treatment has been made
  measured with on the decisional conflict scale. Measured by the decisional conflict scale ( O'Connor, 1995), This contains 16 questions answered on a 5 point likert scale( strongly agree-strongly disagree). Items are given a score value of 0-4. The total score is calculated by: summed, divided by 16 and multiplied by 25. scores range from 0 ( no decisional conflict to 100 (extreme high decisional conflict).
  The scale also consist of 5 subscales: uncertainty subscore, informed subscore, values subscore, support subscore and the effective decision subscore.

SECONDARY OUTCOMES:
Improvement on the perceived level of shared decision making. | 90 days after the decision on their radiation treatment has been made
  measured with the 9-item Shared Decision Making questionnaire (SDM-Q-9,( Kriston 2009)). This contains 9 questions answered on a 6 point likert scale, ranging from 0 ( completely disagree) to 5 ( completely agree). The total score is calculated by: summed score multiplied by 2.2222 transforming to a scale from 0 to 100.
Improvement on the perceived level of shared decision making. | 90 days after the decision on their radiation treatment has been made
  measured with the collaboRATE questionnaire ( Barr 2014), This contains 3 questions answered on a 10 point anchored scale, ranging from 0 ( no effort was made) to 9 ( every effort was made). The total score is calculated by: summed score multiplied by 3.704 transforming to a scale from 0 ( no effort made) to 100 (every effort made).
Patient knowledge | directly after the decision on adjuvant RT has been made (<3 days)
  measured with a ( self developed) knowledge test. This contains 11 questions with 3 possible answers ( True, not true and don't know). For every right answered question 1 point, wrong answers -1 and don't know 0 are given resulting in a range from -11 ( all answers wrong) to 11 ( all answers right).
Decisional conflict | 365 days after the decision on adjuvant RT has been made
  measured with on the decisional conflict scale Measured by the decisional conflict scale ( O'Connor, 1995), This contains 16 questions answered on a 5 point likert scale( strongly agree-strongly disagree). Items are given a score value of 0-4. The total score is calculated by: summed, divided by 16 and multiplied by 25. scores range from 0 ( no decisional conflict to 100 (extreme high decisional conflict).
  The scale also consist of 5 subscales: uncertainty subscore, informed subscore, values subscore, support subscore and the effective decision subscore.
Prospective process evaluation | directly after the decision on adjuvant RT has been made (<3 days)
  how many patients did effectively use the decision aid and how many consultations were needed for the decision to be made. Measured by a log system on the decision aid and by consulting the patients on how many consultations they hade before making the decision.

CONTACTS AND LOCATIONS:
Locations (5):
- Netherlands (5):
  - Radboud UMC, Nijmegen, Gelderland
  - MAASTRO-clinic, Maastricht, Limburg
  - Maastricht University, Maastricht, Limburg
  - Academisch Medisch Centrum (AMC), Amsterdam, North Holland
  - NKI-AVL, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raphael DB, Russell NS, Immink JM, Westhoff PG, Stenfert Kroese MC, Stam MR, van Maurik LM, van den Bongard HJGD, Maduro JH, Sattler MGA, van der Weijden T, Boersma LJ. Risk communication in a patient decision aid for radiotherapy in breast cancer: How to deal with uncertainty? Breast. 2020 Jun;51:105-113. doi: 10.1016/j.breast.2020.04.001. Epub 2020 Apr 6. PMID 32298961